CLINICAL TRIAL: NCT06532318
Title: Comparative Study Between Intralesional Injection of Platelet Rich Plasma and Intralesional Steroid for the Treatment of Trigger Finger in Black Patients
Brief Title: Comparative Study Between Platelet Rich Plasma and Steroid Injection in Trigger Finger Treatment
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Obafemi Awolowo University Teaching Hospital (Other)
Responsible Party: Principal Investigator, Olorunfemi Olayiwola, orthopaedic surgeon, Obafemi Awolowo University Teaching Hospital
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: ERC/2024/06/12
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Trigger Finger Disorder
MeSH Terms: conditions — Trigger Finger Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: All participants will have the same assessment and have blood drawn for CBC. Opaque tape masking of the syringes will be done so that care giver and patients are not aware of interventional drug given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): Patients here will have one milliliter of freshly prepared autologus platelet rich plasma injection for the treatment of their trigger finger.
  Interventions: Biological: Platelet rich plasma
- Group B (Active Comparator): Patients here will have one milliliter(20mg) injection of pfizer Depo-medrol(methylprednisolone acetate) injection for the treatment of their trigger finger.
  Interventions: Drug: Pfizer Depo-medrol

INTERVENTIONS:
Biological: Platelet rich plasma — Freshly prepared autologus platelet rich plasma
  Arms: Group A
Drug: Pfizer Depo-medrol — Methylprednisolone acetate 20mg/ml injection
  Arms: Group B

SUMMARY:
The goal of this clinical trial is to learn if platelet rich plasma works to treat early stage trigger finger in adults. It will also learn about the safety platelet rich plasma. The main questions it aims to answer are:

Does platelet rich plasma lower the pain associated with trigger finger of participants? Does it improve the hand grip strength and Q DASH score of participants? Researchers will compare platelet rich plasma to Depo-Medrol steroid (a known standard of care for early stage trigger finger) to see if platelet rich plasma works to treat early trigger finger.

Participants will:

Take platelet rich plasma or a depo-medrol steroid intralesional injection at recruitment into the intervention Visit the clinic once every 4 weeks for checkups and parameter measurements. Investigator will will keep a record of participants progress in symptom remission

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18year and above with mild or moderate trigger finger, who are willing to have intra-lesional administration of blood product.

No previous treatment for the affected finger.

Exclusion Criteria:

* Previous steroid injection
* Previous Surgery to that finger
* Thrombocytopenic patients
* Hand and finger contracture
* Rheumatoid arthritis of the finger

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-24 (Estimated); Primary Completion 2024-12-23 (Estimated); Study Completion 2025-06-23 (Estimated)

PRIMARY OUTCOMES:
symptom resolution post injection | 3 months
  reduction of pain using VAS and absence snapping of finger

SECONDARY OUTCOMES:
Hand grip strength | 3 month
  measured grip using hand dynamomter
Q- DASH score | 3month
  11-item self reported disability questionnaire that consider upper extremity as one functional unit

IPD SHARING:
Plan to Share IPD: Undecided